CLINICAL TRIAL: NCT06875349
Title: The Effects of Foot Reflexology and Abdominal Massage in Elderly on Constipation: a Randomized Controlled Trial
Brief Title: Foot Reflexology and Abdominal Massage
Acronym: experimental
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Aysun Bayram, assistant professor in nursing fundamentals department, Karadeniz Technical University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2015-KAEK-80-23-30
Record Dates: First submitted 2025-02-20; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Constipation
Keywords: constipation; reflexology; abdominal massage; randomised
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1: Foot Reflexology (Experimental): In the experimental group-1, foot reflexology interventions were applied every three days, with each session lasting 30 minutes, for a total of eight sessions.
  Interventions: Other: foot reflexology
- Group 2: Abdominal Massage (Experimental): In the experimental group-2, abdominal massage interventions were applied every three days, with each session lasting 30 minutes, for a total of eight sessions.
  Interventions: Other: abdominal massage
- Group 3: Control (No Intervention): The elderly individuals in the control group did not receive any intervention and were only monitored.

INTERVENTIONS:
Other: foot reflexology — Foot reflexology is a complementary therapy that involves applying pressure to specific points on the feet, which are believed to correspond to different organs and systems in the body. This technique aims to promote healing by improving blood circulation, reducing stress, and supporting overall well-being. Reflexology is often used to help with issues such as constipation, stress, sleep disorders, and pain management.
  Arms: Group 1: Foot Reflexology
Other: abdominal massage — Abdominal massage is a therapeutic technique that involves applying gentle pressure and circular motions to the abdominal area to stimulate digestion, improve bowel movements, and relieve discomfort. It is commonly used to help with issues such as constipation, bloating, and digestive disorders by promoting intestinal motility and blood circulation. This technique can be performed manually or with the help of tools and is often incorporated into holistic and nursing care practices.
  Arms: Group 2: Abdominal Massage

SUMMARY:
to determine and compare the effects of foot reflexology and abdominal massage applied to elderly individuals on constipation

DETAILED DESCRIPTION:
This randomized controlled study examined the effects of foot reflexology and abdominal massage on constipation in 90 elderly individuals from three nursing homes. Participants were divided into three groups: reflexology, abdominal massage, and control. The intervention groups received eight sessions over three weeks, while the control group received no treatment.

ELIGIBILITY:
Inclusion Criteria:

Being 65 years or older Having no movement restrictions Not using pharmacological laxatives Being diagnosed with constipation according to the ROMA IV criteria Voluntarily agreeing to participate in the study

Exclusion Criteria:

Individuals having a condition that prevents cognitive, affective and verbal communication Having a disorder related to the nervous system and circulatory system Having an injection applied to the abdominal region during the application process Having a systematic disorder related to the GIS (diarrhea, irritable bowel syndrome, fecal impaction, incontinence, etc.) Having physiological and structural disorders that may prevent evacuation in the anus region (rectal fissure, etc.) Having any negativity in the sensory function examination test performed with a sharp-blunt hard object on the sole of the foot and abdomen Having any physiological and structural disorders related to the foot/sole of the foot

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Constipation Severity Scale | Day 1 and Day 13 and Day 25
  Does foot reflexology have an effect on constipation in elderly individuals? Constipation Severity Scale: The total score range is 0-73, with higher scores indicating greater severity of constipation.
Constipation Severity Scale | Day 1 and Day 13 and Day 25
  Does abdominal massage have an effect on constipation in elderly individuals? Constipation Severity Scale: The total score range is 0-73, with higher scores indicating greater severity of constipation.
Constipation Severity Scale | Day 1 and Day 13 and Day 25
  Is there a difference between the effects of foot reflexology and abdominal massage on constipation in elderly individuals? Constipation Severity Scale: The total score range is 0-73, with higher scores indicating greater severity of constipation.

CONTACTS AND LOCATIONS:
Locations (1):
- Karadeniz Technical University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No